CLINICAL TRIAL: NCT06084377
Title: Isolation of Extracellular Embryonic DNA FromIn Vitro Fertilization (IVF) Embryonic Culture Medium and Its Potential Role for Preimplantation Genetic Screening (PGS).
Brief Title: Isolation of Cell Free Fetal DNA From Spent Culture Medium and Its Potential Role for Preimplantation Genetic Diagnosis (PGD).
Status: Completed | Type: Observational
Sponsor: Damascus University (Other)
Responsible Party: Sponsor
Other Study IDs: UDFP-Biochem-01-2023
Record Dates: First submitted 2023-10-11; First posted 2023-10-16 (Actual); Last update posted 2023-10-18 (Actual); Status verified 2023-10

CONDITIONS: Females Undergoing PGD Technology for Medical Conditions
Keywords: Preimplantation Genetic Diagnosis, Spent Culture Medium, cell-free fetal DNA, trophectoderm biopsy

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples With DNA — Spent Culture Medium(SCM)
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Genetic: Preimplantation Genetic Screening — Non-invasive technique to investigate the presence of genetic disorders.
  Other Names: PGS

SUMMARY:
Preimplantation genetic testing for chromosomal screening is, at present, the most reliable method to assess the genetic status of preimplantation embryos. DNA isolated and amplified from trophectoderm (TE) biopsiesis the method currently used for preimplantation genetic testing, but it has significant limitations. There is increasing evidence for a ''true'' noninvasive approach consisting of the analysis of cell-free DNA (cfDNA) released by the embryo into the spent blastocyst medium (SBM) during the late stages of preimplantation development.

This study is to assess whether Noninvasive prenatal genetic diagnosis using cell-free fetal DNA in spent culture medium will substitute for trophectoderm biopsy for heritable disorders screening and if it represents the total fetal genomic DNA.

A total of 27 spent blastocyst media (SBM) from women undergoing IVF will be enrolled with agesless than44 years, whose indications for preimplantation genetic diagnosis for Euploid/Aneuploid embryo determination, were advanced maternal age, recurrent miscarriage, or recurrent implantation failure.We examined the presence of the cell free DNA in spent culture media and whether this DNA is reliable and can be representative of the chromosomal constitution of a blastocyst. So we can affirm that Noninvasive prenatal determination of fetal sex using cell-free fetal DNA (used here as a marker) provides an alternative to invasive techniques for some heritable disorders.

DETAILED DESCRIPTION:
Noninvasiveness is a common theme across medical specialties in the 21st century. In obstetrics, noninvasive prenatal testing provoked a paradigm shift in prenatal clinical practice through the sequencing of fetal cell-free DNA (cfDNA) in maternal plasma. However, current practice for preimplantation genetic testing for aneuploidy (PGT-A) requires trophectoderm biopsy, which entails technical challenges and embryo viability concerns. The possibility to overcome these issues reached the horizon in recent years, with the discovery that cfDNA released by the embryo to the culture media during the latest stages of development offers a new strategy to assess the preimplantation embryo genetically.

Our study evaluates the possibility to isolate fetal cell-free DNA (cfDNA) from culture media and compare the results with TE biopsy samples from the same patients who underwent an IVF stimulation cycle with intracytoplasmic sperm injection at Al-Sharq Hospital between March 2022 and April 2023. During the study's time frame, all embryos were cultured until the blastocyst stage. All enrolled patients underwent niPGD for gender determination using spent culture media as well as standard PGD with TE biopsy using Polymerase chain reaction technique for SRY gene. The embryos were individually cultured in 30-mL media droplets and embryo development progressed using sequential culture media, consistent with routine laboratory practice. For niPGD analysis, the blastocyst-stage culture media on Day 5 was collected (10-20 µl) immediately before TE biopsy was performed. Only embryos achieving a grade 1 (fragmentation less than 15%), were considered eligible for biopsy and vitrification. The embryo culture media samples underwent whole-genome amplification (WGA) using the DOPlify® WGA kit (PerkinElmer) to generate representative amplification of total DNA from spent culture media. The DOP-PCR-based WGA reproducibly amplifies total DNA to produce microgram quantities of amplified and purified genomic DNA in less than 3 hours. We aim to evaluate the concordance rates between trophectoderm biopsy results and cfDNA collected from spent media with an optimized protocol to obtain an adequate quantity and quality of genomic DNA. This interesting work is an important effort to establish the feasibility of the new noninvasive approach that can be a reliable alternative for chromosomal abnormalities assessment of in vitro cultured embryos which will lead to the birth of a living and healthy baby.

Later on, we will perform the SRY gene detection for sex determination using the Polymerase Chain Reaction on the cell-free fetal DNA isolated from spent media samples and compare our results with the TB results.

ELIGIBILITY:
Inclusion Criteria:

* At least two blastocysts suitable for PGD. Only embryos achieving a grade 1 (fragmentation less than 15%).

Exclusion Criteria:

* All embryos do not achieve inclusion criteria as mentioned above.

Ages: 22 Years to 44 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: The study samples will be collected from couples attending Orient Hospital (assisted reproduction and genetics) to carry out the in vitro fertilization process and would like to perform PGD for gender selection. After obtaining the approval of the ethical committee of Damascus University, they will be informed of the research objectives and sign the approve consent.
Sampling Method: Non-Probability Sample
Enrollment: 27 (Actual)
Dates: Start 2020-05-18 (Actual); Primary Completion 2023-04-05 (Actual); Study Completion 2023-09-23 (Actual)

PRIMARY OUTCOMES:
Efficacy of cell free fetal DNA isolated from spent culture medium | At Day 5 of ICSI
  Efficacy of cell free fetal DNA isolated from spent culture medium by Degenerate Oligonucleotide Primed PCR (DOP-PCR)-based Whole Genome Amplification (WGA) for preimplantation genetic analysis.

SECONDARY OUTCOMES:
Increasing the live birth rate, increasing the chances of obtaining embryos free of genetic diseases, and the implantation rate. | 9 Months

CONTACTS AND LOCATIONS:
Overall Officials: Marwan Alhalabi, PhD, Study Chair — Damascus University
Locations (1):
- Damascus University, Damascus, Syria

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Huang J, Rong L, Zeng L, Hu L, Shi J, Cai L, Yao B, Wang XX, Xu Y, Yao Y, Wang Y, Zhao J, Guan Y, Qian W, Hao G, Lu S, Liu P, Qiao J. Embryo selection through non-invasive preimplantation genetic testing with cell-free DNA in spent culture media: a protocol for a multicentre, double-blind, randomised controlled trial. BMJ Open. 2022 Jul 27;12(7):e057254. doi: 10.1136/bmjopen-2021-057254. PMID 35896299
- [Result] Sousa LN, Monteiro PB. Non-invasive preimplantation genetic testing: a literature review. JBRA Assist Reprod. 2022 Aug 4;26(3):554-558. doi: 10.5935/1518-0557.20210102. PMID 35238503
- [Result] Rubio C, Rienzi L, Navarro-Sanchez L, Cimadomo D, Garcia-Pascual CM, Albricci L, Soscia D, Valbuena D, Capalbo A, Ubaldi F, Simon C. Embryonic cell-free DNA versus trophectoderm biopsy for aneuploidy testing: concordance rate and clinical implications. Fertil Steril. 2019 Sep;112(3):510-519. doi: 10.1016/j.fertnstert.2019.04.038. Epub 2019 Jun 11. PMID 31200971
- [Result] Navarro-Sanchez L, Garcia-Pascual C, Rubio C, Simon C. Non-invasive preimplantation genetic testing for aneuploidies: an update. Reprod Biomed Online. 2022 May;44(5):817-828. doi: 10.1016/j.rbmo.2022.01.012. Epub 2022 Jan 31. PMID 35307298
- [Result] Yang L, Lv Q, Chen W, Sun J, Wu Y, Wang Y, Chen X, Chen X, Zhang Z. Presence of embryonic DNA in culture medium. Oncotarget. 2017 Jun 29;8(40):67805-67809. doi: 10.18632/oncotarget.18852. eCollection 2017 Sep 15. PMID 28978073
- [Result] Cornelisse S, Zagers M, Kostova E, Fleischer K, van Wely M, Mastenbroek S. Preimplantation genetic testing for aneuploidies (abnormal number of chromosomes) in in vitro fertilisation. Cochrane Database Syst Rev. 2020 Sep 8;9(9):CD005291. doi: 10.1002/14651858.CD005291.pub3. PMID 32898291
- See also: Related Info — https://pubmed.ncbi.nlm.nih.gov/31200971/
- See also: Related Info — https://pubmed.ncbi.nlm.nih.gov/35307298/
- See also: Related Info — https://www.ncbi.nlm.nih.gov/pmc/articles/PMC9355447/
- See also: Related Info — https://www.ncbi.nlm.nih.gov/pmc/articles/PMC5620213/
- See also: Related Info — https://pubmed.ncbi.nlm.nih.gov/32898291/
- See also: Related Info — https://www.ncbi.nlm.nih.gov/pmc/articles/PMC9335017/